CLINICAL TRIAL: NCT00859144
Title: Community Partnerships to Prevent Urban Youth Health Risks (CHAMPions)
Brief Title: Training Community Members to Deliver HIV Prevention Programs to Urban Youth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCO 03-0888; R01MH069934 (NIH); DAHBR 9A-ASPA
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: HIV; HIV Infections
Keywords: HIV Prevention; Youth; Adolescent; Community Collaboration; Community Mentorship; Minority; Urban; Sexual Risk Behaviors; HIV seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- BART (Experimental): Participants will complete the Becoming a Responsible Teen (BART) program.
  Interventions: Behavioral: Becoming A Responsible Teen (BART)
- Reducing the Risk (Experimental): Participants will complete the Reducing the Risk program.
  Interventions: Behavioral: Reducing the Risk
- Be Proud Be Responsible (Active Comparator): Participants will complete the Be Proud! Be Responsible! program.
  Interventions: Behavioral: Be Proud! Be Responsible!

INTERVENTIONS:
Behavioral: Be Proud! Be Responsible! — This intervention consists of highly structured modules that involve group discussions, videos, games, brainstorming, experiential exercises, and skill building activities. The program encourages participants to be proud of themselves and their community, to behave responsibly for themselves and their community, and to consider their goals for the future and how risk behaviors may interfere with the attainment of their goals.
  Arms: Be Proud Be Responsible
Behavioral: Becoming A Responsible Teen (BART) — This program consists of highly structured modules administered using intervention manuals in community-based settings. Each intervention session involves group discussion, videos, games, presentations, demonstrations, role plays, and practice. Youth learn problem solving, decision-making, communication, condom negotiation and use skills, and behavioral self-management. Youth also meet with HIV infected peers to promote risk recognition and improve their perception of vulnerability.
  Arms: BART
Behavioral: Reducing the Risk — This program consists of instruction on developing social skills to reduce sexual risk-taking behavior and role plays to practice and model skills. Additional activities-such as teaching decision making and assertive communication skills, offering encouragement to obtain relevant health information from stores and clinics, and asking parents about their views on abstinence and birth control-support the premise that students should avoid unprotected intercourse, either by remaining abstinent or using contraceptives.
  Arms: Reducing the Risk

SUMMARY:
This study will examine methods for involving local community members in programs to teach urban youth about how to prevent transmission of HIV.

DETAILED DESCRIPTION:
HIV is a sexually transmitted virus that damages or destroys a body's immune system. When the infection progresses to its later stages, AIDS can develop. Several programs have been developed for educating adolescents about how to prevent HIV transmission. Preventing infection is particularly important because there is not yet a way to cure HIV. This study will examine the processes needed to train community members to deliver HIV prevention programs to urban youth.

This study has three steps. In Step 1, an existing group of urban community members who have already delivered the Be Proud! Be Responsible! HIV prevention program will be invited to serve as mentors for new HIV educators in the community. Participants in this step will complete self-administered assessments of their willingness to collaborate with university-based researchers, their confidence in skills necessary for collaborative projects, and any foreseeable obstacles to participation. The goal of this step is to examine the response over time to ongoing HIV leadership.

In Step 2, parents from the targeted community will be recruited and trained in HIV prevention programs. They will be randomly assigned to one of three programs: Becoming a Responsible Teen, Be Proud! Be Responsible!, and Reducing the Risk. All three of these programs involve group meetings with adolescents to discuss puberty, sexuality, communication, self-esteem, HIV/AIDS, and setting and achieving goals and dreams. Participants in this phase will undergo the same assessments as those in Step 1.

In Step 3, the parents trained in Step 2 will be randomly assigned to a middle school or high school where they will deliver the program in which they were trained. Randomly selected adolescent participants from these schools will be assigned to whichever program is being offered at their school. All three prevention programs will include four to six sessions over 4 to 6 weeks. Adolescent participants will be required to complete interviews and questionnaires when they enter the study, after 3 months, and after 15 months. These interviews and questionnaires will measure HIV/AIDS knowledge, self-esteem, intention to protect health, and engagement in risk-taking behaviors. Parent participants in Step 3 will repeat the assessments from Steps 1 and 2 before and after delivering their prevention curriculums.

ELIGIBILITY:
Inclusion Criteria

* Adult community HIV educators who are parents of a middle or high school aged child
* Adult participants must be between 25 and 60 years of age
* Youth participants must be between 12 and 15 years of age
* Residents of target communities in Bronx, NY

Exclusion Criteria:

* Parent or guardian is excluded if youth participant cannot provide informed consent because of mental health or substance abuse diagnosis
* Significant cognitive impairment that might interfere with understanding of program content or informed consent process

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 901 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Youth sexual risk behaviors | Measured at baseline
  Measured at baseline, after 3 to 4 months, and after 15 months
Youth sexual risk behaviors | Measured after 3 to 4 months
  Measured at baseline, after 3 to 4 months, and after 15 months
Youth sexual risk behaviors | Measured after 15 months
  Measured at baseline, after 3 to 4 months, and after 15 months
HIV educators' intentions to collaborate | Measured at baseline
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
HIV educators' intentions to collaborate | Measured at post-intervention
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
HIV educators' intentions to collaborate | Measured at 3-month follow-up
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
HIV educators' intentions to collaborate | Measured at 15-month follow-up
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
Collaboration by HIV educators | Measured at baseline
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
Collaboration by HIV educators | Measured at post-intervention
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
Collaboration by HIV educators | Measured at 3-month follow-up
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
Collaboration by HIV educators | Measured at 15-month follow-up
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
Youth sexual behavior | Measured at baseline
  Measured at baseline, after 3 to 4 months, and after 15 months
Youth sexual behavior | Measured after 3 to 4 months
  Measured at baseline, after 3 to 4 months, and after 15 months
Youth sexual behavior | Measured after 15 months
  Measured at baseline, after 3 to 4 months, and after 15 months
Youth negotiation of sexual risk situations | Measured at baseline
  Measured at baseline, after 3 to 4 months, and after 15 months
Youth negotiation of sexual risk situations | Measured after 3 to 4 months
  Measured at baseline, after 3 to 4 months, and after 15 months
Youth negotiation of sexual risk situations | Measured after 15 months
  Measured at baseline, after 3 to 4 months, and after 15 months

SECONDARY OUTCOMES:
Leadership skills of HIV educators | Measured at baseline
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
Leadership skills of HIV educators | Measured at post-intervention
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
Leadership skills of HIV educators | Measured at 3-month follow-up
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
Leadership skills of HIV educators | Measured at 15-month follow-up
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
HIV/AIDS knowledge and attitudes of educators and youth | Measured at baseline
  Measured at baseline, after 3 to 4 months, and after 15 months
HIV/AIDS knowledge and attitudes of educators and youth | Measured after 3 to 4 months
  Measured at baseline, after 3 to 4 months, and after 15 months
HIV/AIDS knowledge and attitudes of educators and youth | Measured after 15 months
  Measured at baseline, after 3 to 4 months, and after 15 months
Self-esteem and self-efficacy of HIV educators | Measured at baseline
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
Self-esteem and self-efficacy of HIV educators | Measured at post-intervention
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
Self-esteem and self-efficacy of HIV educators | Measured at 3-month follow-up
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups
Self-esteem and self-efficacy of HIV educators | Measured at 15-month follow-up
  Measured at baseline, post-intervention, and at 3- and 15-month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Mary M. McKay, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States